CLINICAL TRIAL: NCT06784258
Title: Comparison of Inflammatory Factors, Pain Scale, and Postoperative Recovery Quality (QOR - 15) in Patients Undergoing Colorectal Cancer Surgery with Conventional General Anesthesia Techniques Compared to General Anesthesia Combined with Epidural Anesthesia At Prof. Ngoerah Hospital
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Jimmy Wongkar, Medical Doctor, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3005/UN14.2.2.VII.14/LT/2024
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Inflammation Biomarkers; Quality of Recovery (QoR-15); Visual Analog Pain Scale
Keywords: epidural anesthesia; interleukin 6; postoperative pain; colorectal cancer; regional anesthesia; Quality of Recovery-15
MeSH Terms: conditions — Pain, Postoperative; Colorectal Neoplasms | interventions — Anesthesia, General; Control Groups; Anesthesia, Epidural

STUDY DESIGN:
Intervention Model Description: Colorectal patient undergoing elective surgery
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group : Conventinal General Anesthesia (Active Comparator): Patients in the control group will undergo conventional general anesthesia with a regimen of intravenous fentanyl 1-2 mcg/kg body weight, propofol 2-3 mg/kg body weight, and a muscle relaxant for intubation, such as atracurium 0.5 mg/kg body weight or rocuronium 0.6 mg/kg body weight. Afterward, the patient will undergo intubation. Before anesthesia, 2-3 mL of blood will be collected. After the operation is complete the patient will be extubated and blood samples will be taken 6 hours after surgery, VAS (Visual Analog Scale) will be assessed 24 hours postoperatively, and QoR-15 (Quality of Recovery-15) will be evaluated postoperatively. The patient will be given opioid analgesics (Morphine dose 0.5-1 mg/hour given continuously or Fentanyl dose 10-50/hour mcg given continuously), Ketorolac 30 mg every 8 hours intravenously and Paracetamol 500 mg every 6 hours orally
  Interventions: Procedure: General Anesthesia (control group)
- Experimental Group : Conventinal General Anesthesia Combine with Epidural Anesthesia (Experimental): Patients in the experimental group will undergo conventional general anesthesia combine with epidural anesthesia. The patient will undergo epidural anesthesia first with an epidural catheter, the general anesthesia with intravenous fentanyl 1-2 mcg/kg body weight, propofol 2-3 mg/kg body weight, and a muscle relaxant for intubation, such as atracurium 0.5 mg/kg body weight or rocuronium 0.6 mg/kg body weight. Afterward, the patient will undergo intubation. Before anesthesia, 2-3 mL of blood will be collected. After the operation is complete the patient will be extubated and blood samples will be taken 6 hours after surgery, VAS (Visual Analog Scale) will be assessed 24 hours postoperatively, and QoR-15 (Quality of Recovery-15) will be evaluated postoperatively. The patietn will be given Epidural analgesic Bupivacaine 0.1% + Morphine 0.5 mg volume 10 mL every 12 hours, Ketorolac 30 mg every 8 hours + Paracetamol 500 mg every 6 hours orally
  Interventions: Procedure: General Anesthesia combined with epidural anesthesia

INTERVENTIONS:
Procedure: General Anesthesia (control group) — The patient will undergo conventional general anesthesia with a regimen of intravenous fentanyl 1-2 mcg/kg BW, propofol 2-3 ml/kg BW, and muscle relaxants for intubation, such as atracurium 0.5 mg/kg BW or rocuronium 0.6 mg/kg BB. After that the patient will be intubated
  Arms: Control Group : Conventinal General Anesthesia
Procedure: General Anesthesia combined with epidural anesthesia — The patient will undergo epidural anesthesia first with an epidural catheter inserted through a Tuohy needle and ensuring that the length of the multihole epidural catheter that enters the epidural space is 5-6 cm. After that, the patient underwent conventional general anesthesia with a regimen of intravenous fentanyl 1-2 mcg/kg BW, propofol 2-3 ml/kg BW, and muscle relaxants for intubation, such as atracurium 0.5 mg/kg BW or rocuronium 0.6 mg/ kg BW. After that the patient will be intubated. The patient will be given local anesthesia Bupivacaine 0.25% in increments to the desired volume according to the desired height of the segmental block. Local anesthetic medication will be given intermittently every 2 hours
  Arms: Experimental Group : Conventinal General Anesthesia Combine with Epidural Anesthesia

SUMMARY:
Surgery can increase IL-6 cytokines, triggering inflammation and metastasis. The combination of general and epidural anesthesia has the potential to suppress IL-6, improve the tumor microenvironment, provide analgesia, and enhance postoperative recovery.

Objectives :To compare the effectiveness of postoperative analgesia quality in colorectal cancer patients receiving general anesthesia combined with epidural anesthesia.

DETAILED DESCRIPTION:
Patients will be divided into 2 groups: Group P (treatment) and Group K (control).

Before anesthesia, 2-3 mL of blood will be collected by the researcher from patients in both groups using a red tube.

Patients in the control group will undergo conventional general anesthesia. Patients in the treatment group will undergo conventional general anesthesia combined with epidural anesthesia. Patients will be administered 0.25% Bupivacaine local anesthetic incrementally until the desired volume is achieved based on the targeted segmental block height.

Six hours postoperatively, 2-3 mL of blood will be collected, VAS (Visual Analog Scale) will be assessed 24 hours postoperatively, and QoR-15 (Quality of Recovery-15) will be evaluated postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 65 years
* Patients with ASA physical status I - III

Exclusion Criteria:

* Patients with contraindications to regional anesthesia

  * Patients with mental disorders or psychiatric disorders
  * The patient has a history of allergy to the local anesthetic used.
  * The patient or family refuses to take part in the study
  * BMI > 30 Kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-01-28 (Estimated); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
Reduce Interleukin 6 differences | before surgery and 6 hours after surgery
  Interleukin 6 will be collected before surgery and 6 hours after surgery by the anesthesiologist in the Operating theatre.

SECONDARY OUTCOMES:
Reduce VAS pain scale | 24 Hours
  VAS scale will be collected by the anesthesiologist in charge of the patient 24 hours after surgery
Increase Quality of Recovery - 15 | 24 Hours
  QOR-15 score will be collected by the anesthesiologist in charge of the patient 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive Therapy Udayana University, Denpasar, Bali, Indonesia